CLINICAL TRIAL: NCT05695495
Title: Acute Dose-dependent Effects of DMT-bolus Applications in Healthy Subjects: A Placebo-controlled Cross-over Study (DMT BDR-Study).
Brief Title: Acute Dose-dependent Effects of DMT-bolus Applications in Healthy Subjects (DMT BDR-Study)
Acronym: DMT BDR
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: BASEC 2022-01224
Record Dates: First submitted 2022-11-14; First posted 2023-01-25 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Healthy
MeSH Terms: interventions — N,N-Dimethyltryptamine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: In the randomized arm, subjects will be administered intravenous DMT in 4 different bolus doses (5, 10, 15, 20mg) or placebo in randomized, counter-balanced order. In the dose escalation arm, subjects will be administered a placebo and a maximum of 5 DMT bolus doses (5, 10, 15, 20, 25mg) in an escalating dose order. In both arms, the bolus applications will be separated by one hour.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Randomized (Experimental): Subjects will be administered intravenous DMT in 4 different bolus doses or placebo in randomized, counter-balanced order. The bolus applications will be separated by one hour.
  Interventions: Drug: N,N-Dimethyltryptamine (5mg); Drug: N,N-Dimethyltryptamine (10mg); Drug: N,N-Dimethyltryptamine (15mg); Drug: N,N-Dimethyltryptamine (20mg); Drug: Placebo (saline)
- Dose ecalation (Experimental): Subjects will be administered a placebo and a maximum of 5 DMT bolus doses in an escalating dose order. The bolus applications will be separated by one hour.
  Interventions: Drug: N,N-Dimethyltryptamine (5mg); Drug: N,N-Dimethyltryptamine (10mg); Drug: N,N-Dimethyltryptamine (15mg); Drug: N,N-Dimethyltryptamine (20mg); Drug: N,N-Dimethyltryptamine (25mg); Drug: Placebo (saline)

INTERVENTIONS:
Drug: N,N-Dimethyltryptamine (5mg) — Intravenous bolus application over 45 seconds
Drug: N,N-Dimethyltryptamine (10mg) — Intravenous bolus application over 45 seconds
Drug: N,N-Dimethyltryptamine (15mg) — Intravenous bolus application over 45 seconds
Drug: N,N-Dimethyltryptamine (20mg) — Intravenous bolus application over 45 seconds
Drug: N,N-Dimethyltryptamine (25mg) — Intravenous bolus application over 45 seconds
  Arms: Dose ecalation
Drug: Placebo (saline) — Intravenous bolus application over 45 seconds

SUMMARY:
N,N-dimethyltryptamine (DMT) is a psychoactive substance with similar effects such as LSD or psilocybin. However, DMT is less well characterized than the latter substances. The present study is a modern randomized cross-over trial, investigating different intravenous DMT boluses over a broad dose range. Thus, different doses will be tested and related to subjective and autonomic effects.

DETAILED DESCRIPTION:
N,N-dimethyltryptamine (DMT) is a naturally-occurring psychedelic substance widely used in recreational and spiritual settings (Ayahuasca). DMT is considered a tool to induce an altered state of consciousness of interest in psychological and psychiatric research. DMT is rapidly metabolized by monoamine oxidase (MAO) A. Therefore, it is inactive when administered orally and has a very short duration of action when administered parenterally (<20 min). However, to date no clinical study has investigated dose-response effects over a broad range of different doses of DMT within the same patient. The aim of the present study is to experimentally test different intravenous DMT bolus doses over a broad dose range and investigate the related subjective and autonomic effects in order to establish a precise dose-response relationship of DMT in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 25 and 65 years old
2. Sufficient understanding of the German language
3. Understanding of procedures and risks associated with the study
4. Willing to adhere to the protocol and signing of the consent form
5. Willing to refrain from the consumption of illicit psychoactive substances during the study
6. Abstaining from xanthine-based liquids from the evenings prior to the study sessions and during the sessions
7. Willing not to operate heavy machinery within 6 h of DMT administration
8. Willing to use double-barrier birth control throughout study participation
9. Body mass index between 18-29 kg/m2.

Exclusion Criteria:

1. Chronic or acute medical condition
2. Current or previous major psychiatric disorder (e.g. psychotic disorders, mania / hypomania, anxiety disorders).
3. Psychotic disorder or bipolar disorder in first-degree relatives
4. Hypertension (SBP>140/90 mmHg) or hypotension (SBP<85 mmHg)
5. Hallucinogenic substance use (not including cannabis) more than 20 times or any time within the previous two months
6. Pregnancy or current breastfeeding
7. Participation in another clinical trial (currently or within the last 30 days)
8. Use of medication that may interfere with the effects of the study medication
9. Tobacco smoking (>10 cigarettes/day)
10. Consumption of alcoholic beverages (>20 drinks/week)

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2024-06-12 (Actual); Primary Completion 2025-02-02 (Actual); Study Completion 2025-03-04 (Actual)

PRIMARY OUTCOMES:
Altered states of consciousness profile (OAV) | Repeatedly 1 hour after each bolus application
  Altered states of consciousness profile (OAV) consisting of 42 items to be rated on a visual analog scale (0-100 mm), with higher values indicating stronger effects with higher scores representing more intense effects
Subjective effect ratings over time | Repeatedly 1 hour after each bolus application
  Participants will be asked by the investigator to repeatedly rate their subjective effects verbally on a Likert scale from 0 to 10 for: "any drug effect", "good drug effect", "bad drug effect", and "fear". Ratings will be performed before and repeatedly after substance administration and will take approximately 30 sec complete.

SECONDARY OUTCOMES:
Psychedelic experience questionnnaire (PEQ) | Repeatedly 1 hour after each bolus application
  Assesses the emergence and intensity of phenomenons occurring in altered states of consciousness on a 6-point Likert scale ranging from 0 ("not at all") to 5 ("extremely").
Near death experience content scale (NDE-C) | Repeatedly 1 hour after each bolus application
  The Near-Death Experience Content (NDE-C) scale is a tool to assess dimensions of near-death experience on a Likert scale ranging from 0 ("not at all") to 4 ("extremely").
Spiritual Realms Questionnaire (SRQ) | Once at the end of study day
  Assesses the spiritual phenomenons elicited by psychedelic substances through 11 main questions to be answered on a total of 65 sub-ordered 100mm visual analog scales once on each study day
Blood pressure | Repeatedly in short intervals (2-10 minutes) after each bolus application
  Assessed multiple times on each study day via systolic and diastolic blood pressure
Heart rate | Repeatedly in short intervals (2-10 minutes) after each bolus application
  Assessed multiple times on each study day.
Plasma level DMT | Repeatedly in short intervals (2-10 minutes) after each bolus application
  Assessed multiple times on each study day.
Urine recovery of DMT | Once at the end of study day
  Assessed once on each study day
NEO-Five-Factor-Inventory (NEO-FFI) | Baseline
  The NEO-FFI is a self-description questionnaire with 60 items for the measurement of the "big five": neuroticism, extraversion, openness, agreeableness, and consciousness. It uses a 5-point Likert scale ranging from "completely disagree" to "fully agree.
Saarbrücker Personality Questionnaire (SPF) | Baseline
  The SPF defines empathy as the "reactions of one individual to the observed experiences of another." It assesses 28- items on a 5-point Likert scale ranging from "Does not describe me well" to "Describes me very well". The measure has 4 subscales (Perspective Taking, Fantasy, Empathic Concern, Personal Distress) each made up of 7 different items.
Elliot Humility Scale (EHS) | Baseline
  The Elliot Humility Scale (EHS) is a validated 13-item self-rating measure assessing four subscales, i.e. openness, self-forgetfulness, accurate self-assessment, and focus on others on a 5-point Likert scale ranging from "strongly disagree" to "strongly agree"

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Pharmacology & Toxicology, University Hospital Basel, Basel, Switzerland